CLINICAL TRIAL: NCT04133688
Title: A Mobile App for the Self Quantification of Sleep and Behaviors : a Pilot Study With Teenagers and Young Adults
Brief Title: Mobile App in Addiction
Acronym: ASC-Val
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-A01374-51
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Addiction
Keywords: mobile app, pilot study, addiction, sleep, ePRO
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application (ASC) (Experimental): mobile app / devise
  Interventions: Device: ASC
- Paper diary (Active Comparator): paper diary
  Interventions: Device: ASC

INTERVENTIONS:
Device: ASC — mobile app
  Other Names: mobile application

SUMMARY:
The sleep and behavior agendas are today very largely underused while they can be of a considerable contribution in the follow-up of the patients and the reinforcement of the therapeutic alliance. In the management of addictions, sleep disorders are a major comorbidity, these two components maintain indeed complex links: it was highlighted a bidirectional relationship between the effect of the consumption of addictive substances on sleep and conversely, the effect of sleep disorders on the consumption of products, the same is true for overexposure to screens.

DETAILED DESCRIPTION:
The sleep and behavior agendas are today very largely underused while they can be of a considerable contribution in the follow-up of the patients and the reinforcement of the therapeutic alliance. In the management of addictions, sleep disorders are a major comorbidity, these two components maintain indeed complex links: it was highlighted a bidirectional relationship between the effect of the consumption of addictive substances on sleep and conversely, the effect of sleep disorders on the consumption of products, the same is true for overexposure to screens.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers or young adults from 12 to 18 years old (included)
* Consultant for addiction to cannabis and / or tobacco and / or alcohol and / or screen
* Treated within the Functional Unit of addictology
* For minors, after parental consent

Exclusion Criteria:

-

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Number of days filled for sleep and consumptions, usable by the doctor on the day of the consultation / after 15 days of self-evaluation required by the treatment | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Pitrat, MD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France